CLINICAL TRIAL: NCT03419871
Title: Sleep, Biological Stress, and Health Among Toddlers Living in Socioeconomically Disadvantaged Homes
Brief Title: Associations of Socioeconomic Adversity and Sleep With Allostatic Load Among Toddlers
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1504015764
Record Dates: First submitted 2017-12-19; First posted 2018-02-05 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Sleep Disorder
Keywords: economically stressed communities
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- monitoring sleep effects on toddlers: Monitoring the sleep characteristics of toddlers living in economically stressed communities.
  Interventions: Other: Monitoring Sleep; Other: stress biomarkers

INTERVENTIONS:
Other: Monitoring Sleep — An accelerometer will be placed on the wrist or ankle of the child while the child sleeps in their home. Caregivers will be instructed to keep the accelerometer on their toddler's ankle to measure sleep duration, latency and sleep efficiency. Seven nights of data will be obtained because actigraphy is most reliably measured in young children over this time frame.
Other: stress biomarkers — Salivary and hair cortisol measurements were used to obtain a change in baseline from 12 to 24 months. Data on the timing of the saliva collection will be collected using a Medical Electronic Monitoring System (MEMScapTM) - a digital memory cap that records the timing and frequency of opening.
  Cortisol will be measure in the morning and bedtime samples. A small amount of hair (30mg) will be cut from the posterior vertex of the child's head. Due to the expected variability in hair length of toddlers, documentation of hair length will be completed. Each centimeter represents 1 month history of stress and ideally 3 cm of hair length will be collected to provide a three month history of stress.

SUMMARY:
A longitudinal study to examine the relationships among sleep characteristics, stress, and child behavior problems in a community sample of toddlers (12-24 months- ages 12-15 months at enrollment) living in socioeconomically disadvantaged homes

DETAILED DESCRIPTION:
The purpose of this study is to examine the relationships among sleep characteristics, stress (allostatic load), and health among toddlers living in economically stressed communities. Sleep difficulty, including short sleep duration and poor sleep efficiency, is closely related to measures of stress, including interleukin (IL-6), cortisol, c-reactive proteins (CRP), secretory immunoglobulin A (SIgA), and body mass index (BMI) and may therefore contribute to 'wear and tear' on the body (allostatic load), a problem that places children at high risk of physical and mental health problems. Young children who live with socioeconomic adversity are especially vulnerable to both sleep difficulty and higher levels of physiologic stress (allostatic load).

ELIGIBILITY:
Inclusion Criteria:

* Toddlers (12-24 months- ages 12-15 months at enrollment) living in socioeconomically disadvantaged homes.

Exclusion Criteria:

* If the toddler has a diagnosis of sleep apnea or has another documented medical condition affecting sleep.

Ages: 12 Months to 15 Months | Sex: All
Age Groups: Child
Study Population: Toddlers (12-24 months- ages 12-15 months at enrollment) living in socioeconomically disadvantaged homes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11-08 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Sleep monitoring | 9 days
  Sleep characteristics will be measured by an accelerometer on the wrist or ankle to measure sleep efficiency.
Caregiver report | 12 to 36 months
  Caregivers will complete the Brief Infant Sleep Questionnaire
Sleep diary | 12 to 24 months
  Caregivers will complete a sleep diary to record their toddler's sleep for time period when an accelerometer will be worn by the child.
Behavioral monitoring | 12 to 36 months
  Toddler behavior problems will be assessed using the Brief Infant Toddler Social and Emotional Assessment (BITSEA).

SECONDARY OUTCOMES:
Cortisol biomarker | 12 to 24 months
  A small amount of hair (30mg) will be cut from the posterior vertex of the child's head. The samples will be tied together with the scalp end noted.
Immune biomarkers | 12 to 24 months
  A secretory antibody immunoglobulins A and secretory immunoglobulins A ( IgA ,S-IgA) that plays an integral role in the maintenance of mucosal homeostasis and is associated with increased risk of infection will be measured.
Anthropometric biomarkers | 12 to 24 months
  Anthropometrics - Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ordway, Phd, Principal Investigator — Yale University School of Nursing
Locations (1):
- Yale New Haven Hospital Primary Care Center, New Haven, Connecticut, United States